CLINICAL TRIAL: NCT04618757
Title: Trial Evaluating Hedonic vs Cash Incentives
Acronym: TEH-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NIHA-2018-002 (Study 1)
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hedonic Reward (Experimental): Participants' reward for meeting monthly step targets is in the form of reimbursements of up to $50 for expenses on hedonic activities of their choice
  Interventions: Behavioral: Hedonic Reward; Device: Fitbit
- Cash Reward (Experimental): Participants' reward for meeting monthly step targets is in the form of $50 cash disbursements
  Interventions: Behavioral: Cash Reward; Device: Fitbit

INTERVENTIONS:
Behavioral: Hedonic Reward — A reimbursement credit for hedonic expenses worth up to $50 will be awarded to each participant if they log at least 10,000 daily steps on at least 25 days during the first 28 days of each calendar month on Fitbit activity trackers provided by the study.
  Arms: Hedonic Reward
Behavioral: Cash Reward — A reimbursement credit for $50 in cash will be awarded to each participant if they log at least 10,000 daily steps on at least 25 days during the first 28 days of each calendar month on Fitbit activity trackers provided by the study.
  Arms: Cash Reward
Device: Fitbit — Fitbit devices are wireless pedometers that track the steps of participants, and will be offered in conjunction with a tailored website with customized information for participants.
  Other Names: Fitbit, wireless pedometer, physical activity tracker

SUMMARY:
This study aims to determine, using a randomized trial with two parallel arms, whether hedonic rewards (Arm 1) can be more effective than their cash equivalent (Arm 2) in motivating participants to meet step goals.

DETAILED DESCRIPTION:
The evidence is overwhelming that sustained physical activity reduces risks for non-communicable diseases, increases longevity, and reduces medical costs. Yet, the rates of physical activity have been steadily decreasing such that physical inactivity is now the fourth leading cause of death worldwide. In Singapore, 33% of adults are insufficiently active despite Singapore being a highly walkable city with numerous subsidized community-based physical activity programs. A review of the literature shows that, to date, no study has directly compared cash versus hedonic rewards for health behavior change despite theory suggesting hedonic rewards may work better. Furthermore, hedonic rewards can often be purchased at lower cost than their cash equivalent. This makes hedonic rewards potentially more cost-effective if they are proven to be at least as effective at increasing positive behavior change compared to giving the same value in cash.

Thus, we aim to determine, using a randomized trial with two parallel arms, whether hedonic rewards (Arm 1) can be more effective than their cash equivalent (Arm 2) in promoting increases in physical activity, assessed via step counts measured by a Fitbit physical activity tracker, during a 4-calendar month intervention. We hypothesize that the average proportion of months meeting the incentivized step target across participants will be greater for those in the hedonic incentive arm as compared to those in the cash incentive arm (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 to 70 years inclusive.
* Singapore resident (residing in Singapore during the study period [up to 5 months])
* English-speaking and English literate
* Smartphone-literate

Exclusion Criteria:

* Pregnant or lactating
* Unable to walk up 10 steps (individual steps, not floors) without stopping
* Currently on doctor's advice against engaging in moderate-to-vigorous physical activity (i.e., brisk walking or more intense).
* Currently have a condition(s) that restricts engaging in moderate-to-vigorous physical activity (i.e., brisk walking or more intense).
* Unwilling to be randomized into study arms
* Unwilling to use a Fitbit for the study period (up to 5 calendar months)
* Unwilling to pay the $20 enrolment fee
* Does not complete the Consent Form
* Refuses to give consent to participate in the study

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of months in meeting the step target | Months 1-4
  The mean proportion of months meeting the incentivized targets (i.e. at least 10,000 daily steps on at least 25 days during the first 28 days of each calendar month via step counts measured by Fitbit, during a 4 calendar month intervention) across participants.

SECONDARY OUTCOMES:
Difference in mean daily steps between the 2 intervention arms | Months 1-4
  Difference in mean daily steps between intervention arms for the first 28 days of each of 4 intervention months, controlling for baseline daily values. These will be measured via step counts measured by Fitbit.
Difference in median daily steps between the 2 intervention arms | Months 1-4
  Difference in median daily steps between intervention arms for the first 28 days of each of 4 intervention months, controlling for baseline daily values. These will be measured via step counts measured by Fitbit.
Difference in mean Fitbit fairly and very active minutes between the 2 intervention arms | Months 1-4
  Difference in mean Fitbit fairly and very active minutes between intervention arms for the first 28 days of each of 4 intervention months, controlling for baseline daily values. The Fitbit fairly and active minutes count towards Fitbit "active minutes", which are determined by Fitbit's proprietary algorithms and are defined as sustained activity of ≥10-minute bouts. These will be measured via step counts measured by Fitbit.
Difference in median Fitbit fairly and very active minutes between the 2 intervention arms | Months 1-4
  Difference in median Fitbit fairly and very active minutes between intervention arms for the first 28 days of each of 4 intervention months, controlling for baseline daily values. The Fitbit fairly and active minutes count towards Fitbit "active minutes", which are determined by Fitbit's proprietary algorithms and are defined as sustained activity of ≥10-minute bouts. These will be measured via step counts measured by Fitbit

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, Ph.D, M.H.A, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Medical School, Singapore, Singapore

REFERENCES:
- [Derived] Finkelstein EA, Chow MTN, Gandhi M. Are cash incentives always king? A randomized controlled trial evaluating hedonic versus cash incentives (TEH-C). Front Public Health. 2024 Apr 30;12:1354814. doi: 10.3389/fpubh.2024.1354814. eCollection 2024. PMID 38745998